CLINICAL TRIAL: NCT06622512
Title: Double-Blind Randomized Controlled Trial Comparing the Effectiveness of Two Standardized Radial Pressure Wave Techniques Versus Pain-Site Guided Therapy in Patients With Knee Osteoarthritis.
Brief Title: Two Standardized Radial Pressure Wave Techniques Versus Pain-Site Guided Therapy in Patients With Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Armando Tonatiuh Avila Garcia, Chief Department of Physical Medicine and Rehabilitation, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI 157/24
Record Dates: First submitted 2024-09-20; First posted 2024-10-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; osteoarthritis; extracorporeal shock wave therapy; radial pressure wave therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomization After having obtained written informed consent the patients will be randomly assigned to one of three treatment groups, RPWT at the two most painful points (control group), RPWT at the medial interarticular line (medial group) or RPWT at the medial and lateral interarticular lines (medial and lateral group). Randomization will be carried out using the paper envelope randomization method. For this purpose, we will prepare a series of opaque papers, each indication one of the three possible assignments. These papers will be placed in an opaque bag, and during the enrollment process, each patient will draw a paper from the bag at random. The patient´s group assignment will be determined by the designation on the drawn paper.
Who Masked: Participant, Investigator
Masking Description: Blinding This study will employ a double-blind design, in which both the participants and the clinical evaluator responsible for conducting clinical and radiographic assessments will be blinded to the group assignments. Participants will be informed that they may receive one of three possible treatment options but will not know which specific technique is being applied to them. The RPWT will be administered by a final-year resident physician in Physical Medicine and Rehabilitation, who will be aware of the group allocation but will have no involvement in the outcome assessments. To ensure further blinding, the data collection and analysis personnel will also be blinded to the intervention groups. All treatment sessions will be conducted under standardized conditions, with identical instructions, setup, and environment for all groups to reduce potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): The three groups will receive RPWT with the device BTL-6000 Radial Shockwave Therapy (BTL Industries, Ltd.). Each patient, in supine position and knee flexion of 30 to 60 degrees, will receive 3 sessions of RPW, once per week, 2,000 impulses per session, 2.0 bar and frequency of 10Hz. The air pressure and frequency will be adjusted in response to discomfort. The control group will receive 1,000 pulses at the two most painful sites of the treated knee, in accordance with the technique employed in the majority of previous studies in this field.
  Interventions: Device: Radial Pressure Wave Therapy
- Medial group (Experimental): The three groups will receive RPWT with the device BTL-6000 Radial Shockwave Therapy (BTL Industries, Ltd.). Each patient, in supine position and knee flexion of 30 to 60 degrees, will receive 3 sessions of RPW, once per week, 2,000 impulses per session, 2.0 bar and frequency of 10Hz. The air pressure and frequency will be adjusted in response to discomfort. The medial group will receive 2,000 pulses at the medial interarticular line of the treated knee.
  Interventions: Device: Radial Pressure Wave Therapy
- Medial and lateral group (Experimental): The three groups will receive RPWT with the device BTL-6000 Radial Shockwave Therapy (BTL Industries, Ltd.). Each patient, in supine position and knee flexion of 30 to 60 degrees, will receive 3 sessions of RPW, once per week, 2,000 impulses per session, 2.0 bar and frequency of 10Hz. The air pressure and frequency will be adjusted in response to discomfort. The medial and lateral group will receive 1,000 pulses at the medial interarticular line and 1,000 pulses at the lateral interarticular line of the treated knee.
  Interventions: Device: Radial Pressure Wave Therapy

INTERVENTIONS:
Device: Radial Pressure Wave Therapy — Radial pressure wave therapy (RPWT) is a non-invasive treatment used for musculoskeletal disorders, including knee OA. (Schroeder AN) It involves the application of mechanical energy to stimulate biological responses, RPWT differs fundamentally from focal shock wave therapy (FSWT) in several physical properties, in its point of maximum energy flux density (EFD), and in some clinical applications. RPWT activates cellular pathways involved in tissue regeneration and generates mechanical energy that spreads radially from the point of application, primarily affecting superficial tissues and leading to pain relief and improved function through a process known as mechano-transduction, by enhancing blood flow and stimulating cellular repair processes . (Simplicio CL, Wang CJ)

SUMMARY:
The goal of this clinical trial is to evaluate and compare the effectiveness of radial pressure wave therapy (RPWT) applied at different anatomical sites in patients with knee osteoarthritis (OA) over a follow-up of four months. The main questions it aims to answer are:

How effective is the application of RPWT on the medial and lateral interarticular lines in patients with knee OA? Are standardized RPWT application techniques on interarticular lines superior to the traditional application technique on the points of greatest pain in patients with knee OA?

Researchers will compare the effectiveness of two standardized application techniques on interarticular lines to decrease pain and improve function in patients with knee OA.

Participants will receive three sessions of RPWT on the most painful knee as a result of knee OA.

DETAILED DESCRIPTION:
Methods Patients The study will enroll patients between the ages of 50 and 80 years with chronic and current knee pain and a clinical and radiographic diagnosis of knee osteoarthritis (OA). Participants will be recruited through the "Treatment of Knee OA with Radial Pressure Wave Therapy" campaign conducted by the Physical Medicine and Rehabilitation Department of the Hospital Civil de Guadalajara "Fray Antonio Alcalde" in México. Recruitment will take place during the months of August and September 2024. Individuals with a history of knee surgery, inflammatory arthritis, septic arthritis, fibromyalgia, cancer, or severe vascular insufficiency will be excluded from participation in this study.

Ethical Statement The participants will be required to sign an informed consent form which will include all details of the study. The patients will be free to decide whether or not to participate or to withdraw from the protocol at any time. The study was approved by the Research Ethics Committee of the Hospital Civil de Guadalajara Fray Antonio Alcalde (number: CEI 157/24) and was conducted in accordance with the World Medical Association's Declaration of Helsinki.

Randomization After obtaining written informed consent, the participants will be randomized to one of three treatment groups: radial pressure wave therapy (RPWT) at the two most painful points (control group), RPWT at the medial interarticular line (medial group), or RPWT at the medial and lateral interarticular lines (medial and lateral group). Randomization will be performed using the paper envelope randomization method. For this purpose, the investigators will prepare a series of opaque papers, each indicating one of the three possible assignments. These papers will be placed in an opaque bag, and during the enrollment process, each patient will randomly draw a paper from the bag. The patient's group assignment will be determined by the label on the paper drawn.

Treatment The three groups will receive RPWT using the BTL-6000 Radial Shockwave Therapy device (BTL Industries, Ltd.). Each patient will receive 3 sessions of RPW, once a week, in the supine position with knee flexion of 30 to 60 degrees, 2,000 pulses per session, 2.0 bar, and frequency of 10 Hz. The air pressure and frequency will be adjusted according to discomfort. The control group will receive 1,000 pulses to the two most painful areas of the treated knee, according to the technique used in most previous studies in this area. The medial group will receive 2,000 pulses at the medial interarticular line of the treated knee, while the medial and lateral groups will receive 1,000 pulses at the medial interarticular line and 1,000 pulses at the lateral interarticular line of the treated knee. All participants will be trained to perform a home exercise program for 4 consecutive weeks, three sessions per week, consisting of superficial thermotherapy for 10 minutes, hamstring and quadriceps stretching, medial gluteus medius and quadriceps strengthening, and propioception exercises. The interventions will be performed at the Physical Medicine and Rehabilitation Department of the Civil Hospital of Guadalajara "Fray Antonio Alalde". Complications, adverse effects and complaints during treatment will be documented.

Outcome measures A questionnaire will be used to assess sociodemographic characteristics, including age, gender, and education level for all patients. In addition, the numerical and categorical forms of body mass index (BMI), physical activity habits, and analgesic use will be assessed after eligibility criteria are established using the aforementioned instrument. The severity of knee OA will also be measured by a board-certified rheumatologist using the Kellgren & Lawrence scale.

The Spanish version of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be used to assess self-reported disability. The WOMAC is a disease-specific, self-administered questionnaire developed for patients with knee OA and takes approximately 5 minutes to complete. It has a multidimensional scale consisting of 24 items grouped into three dimensions: pain (five items), stiffness (two items), and physical function (17 items). We will use the Likert version with five response levels for each item, representing different levels of intensity (none, mild, moderate, severe or extreme) that are scored from 0 to 4. The final score for the WOMAC questionnaire is determined by adding the aggregate scores for pain, stiffness and function. The higher the score, the worse the patient's condition; therefore, improvement is achieved by reducing the total score. The data were standardized to a range of 0 to 100, with 0 representing the best possible health status and 100 representing the worst possible status. Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), a world-renowned instrument consisting of a linear scale with numbered intervals from zero (no pain) to ten (the worst pain) that patients use to quantify their current pain intensity. It is well known that pain is the most important symptom of knee OA. Therefore, pain will be the primary outcome measure in the study. Treatment success was defined as an individual improvement in the NPRS of 50% from baseline. Evaluations will be performed at baseline, at the end of the third session, at 2 months, and at 4 months after the first RPWT session.

Blinding This study will use a double-blind design in which both the participants and the clinical evaluator responsible for performing the clinical and radiographic assessments will be blinded to the group assignments. Participants will be informed that they may receive one of the three possible treatment options, but will not know which specific technique will be applied to them. The RPWT will be performed by a final year resident in Physical Medicine and Rehabilitation who will be aware of the group assignments but will not be involved in the outcome assessments. To ensure further blinding, data collection and analysis personnel will also be blinded to the intervention groups. All treatment sessions will be conducted under standardized conditions with identical instructions, setup, and environment for all groups to reduce potential bias.

Sample size calculation Pain intensity, as measured by the NPRS, was considered the primary outcome measure for sample size determination. The investigators used a significance level of 0.05 (two-tailed) and statistical power of 80% (1-β), corresponding to Z values of 1.96 and 0.84, respectively. The calculation was based on an expected effect size of 2.0, considered clinically relevant based on previous studies, and a standard deviation of 2.1 reported in the literature. The initial calculation indicated that approximately 17 participants per group would be required. To account for an expected 20% loss to follow-up, the investigators adjusted the sample size and increased it to 23 participants per group to ensure the robustness and validity of the results. In summary, a total of 23 patients will be recruited for each of the three groups in our study, taking into account both the expected effect size and the adjustment for loss to follow-up.

Statistical Analysis Data will be analyzed using the Statistical Package for the Social Sciences (SPSS) version 22.0 software. Normality of the data distribution was assessed using the Kolmogorov-Smirnov test. For variables with a normal distribution, the mean and standard deviation will be calculated; for variables with a non-normal distribution, the median and interquartile range (IQR) will be reported. Qualitative data are presented as numbers and percentages. In cases of normal distribution, a t-test will be used to analyze differences within and between groups. One-way ANOVA will be used to determine statistical differences in WOMAC questionnaire and NPRS scores over the course of the study. Pearson's correlation coefficient will be used to assess the relationship between the 4th month scores (WOMAC and NPRS), baseline scores, age, BMI, and Kellgren & Lawrence severity grades. The strength of the correlation is classified as negligible (0.00-0.10), weak (0.10-0.39), moderate (0.40-0.69), strong (0.70-0.89), and very strong (0.90-1.00). All tests are considered statistically significant at a p-value of ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Chronic and current knee pain.
* Clinical and radiographic diagnosis of knee OA.

Exclusion Criteria:

* History of knee surgery.
* Inflammatory arthropathy.
* Septic arthritis.
* Fibromyalgia.
* Cancer.
* Severe vascular insufficiency

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | At baseline, at the end of the third session, two months after the first session, and four months after the first session.
  Pain intensity will be assessed using the Numeric Pain Rating Scale, a world-renowned instrument consisting of a linear scale with numbered intervals from zero (no pain) to ten (the worst pain) that patients use to quantify their current pain intensity.
Self-reported disability | At baseline, at the end of the third session, two months after the first session, and four months after the first session.
  Self-reported disability measured with the Western Ontario and McMaster Universities Osteoarthritis Index, a disease-specific, self-administered questionnaire developed for patients with knee osteoarthritis and takes approximately 5 minutes to complete. It has a multidimensional scale consisting of 24 items grouped into three dimensions: pain (five items), stiffness (two items), and physical function (17 items). We will use the Likert version with five response levels for each item, representing different levels of intensity (none, mild, moderate, severe or extreme) that are scored from 0 to 4. The final score for the questionnaire is determined by adding the aggregate scores for pain, stiffness and function. The higher the score, the worse the patient's condition; therefore, improvement is achieved by reducing the total score. The data were standardized to a range of 0 to 100, with 0 representing the best possible health status and 100 representing the worst possible status.

CONTACTS AND LOCATIONS:
Overall Officials: Tonatiuh Avila, MD, Principal Investigator — Hospital Civil de Guadalajara
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study are available from the lead author upon reasonable request by email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From February 2025 to February 2026.
Access Criteria: 1. Qualified researchers who have received IRB approval.
  2. Prior reasonable request by email.
  3. Data will be made available by PDF files or other non-editable formats.

REFERENCES:
- [Background] O'Neill TW, Felson DT. Mechanisms of Osteoarthritis (OA) Pain. Curr Osteoporos Rep. 2018 Oct;16(5):611-616. doi: 10.1007/s11914-018-0477-1. PMID 30155845
- [Background] Giorgino R, Albano D, Fusco S, Peretti GM, Mangiavini L, Messina C. Knee Osteoarthritis: Epidemiology, Pathogenesis, and Mesenchymal Stem Cells: What Else Is New? An Update. Int J Mol Sci. 2023 Mar 29;24(7):6405. doi: 10.3390/ijms24076405. PMID 37047377
- [Background] Primorac D, Molnar V, Rod E, Jelec Z, Cukelj F, Matisic V, Vrdoljak T, Hudetz D, Hajsok H, Boric I. Knee Osteoarthritis: A Review of Pathogenesis and State-Of-The-Art Non-Operative Therapeutic Considerations. Genes (Basel). 2020 Jul 26;11(8):854. doi: 10.3390/genes11080854. PMID 32722615
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Geng R, Li J, Yu C, Zhang C, Chen F, Chen J, Ni H, Wang J, Kang K, Wei Z, Xu Y, Jin T. Knee osteoarthritis: Current status and research progress in treatment (Review). Exp Ther Med. 2023 Aug 25;26(4):481. doi: 10.3892/etm.2023.12180. eCollection 2023 Oct. PMID 37745043
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Allaeys C, Arnout N, Van Onsem S, Govaers K, Victor J. Conservative treatment of knee osteoarthritis. Acta Orthop Belg. 2020 Sep;86(3):412-421. PMID 33581025
- [Background] De la Corte-Rodriguez H, Roman-Belmonte JM, Rodriguez-Damiani BA, Vazquez-Sasot A, Rodriguez-Merchan EC. Extracorporeal Shock Wave Therapy for the Treatment of Musculoskeletal Pain: A Narrative Review. Healthcare (Basel). 2023 Oct 26;11(21):2830. doi: 10.3390/healthcare11212830. PMID 37957975
- [Background] Zhou Q, Chen J. A critical overview of systematic reviews and meta-analyses of extracorporeal shockwave therapy for knee osteoarthritis. Asian J Surg. 2024 Jul;47(7):2975-2984. doi: 10.1016/j.asjsur.2024.01.127. Epub 2024 Jan 30. PMID 38290944
- [Background] Imamura M, Alamino S, Hsing WT, Alfieri FM, Schmitz C, Battistella LR. Radial extracorporeal shock wave therapy for disabling pain due to severe primary knee osteoarthritis. J Rehabil Med. 2017 Jan 19;49(1):54-62. doi: 10.2340/16501977-2148. PMID 27904912
- [Background] Tornese D, Mattei E, Lucchesi G, Bandi M, Ricci G, Melegati G. Comparison of two extracorporeal shock wave therapy techniques for the treatment of painful subcalcaneal spur. A randomized controlled study. Clin Rehabil. 2008 Sep;22(9):780-7. doi: 10.1177/0269215508092819. PMID 18728131
- [Background] Zhang YF, Liu Y, Chou SW, Weng H. Dose-related effects of radial extracorporeal shock wave therapy for knee osteoarthritis: A randomized controlled trial. J Rehabil Med. 2021 Jan 13;53(1):jrm00144. doi: 10.2340/16501977-2782. PMID 33367924